CLINICAL TRIAL: NCT04717115
Title: An International Study on Genotype/Phenotype Correlation With Focus on Lung Function in Patients With Primary Ciliary Dyskinesia (PCD)
Brief Title: Genotype/Phenotype Correlation With Focus on Lung Function in Primary Ciliary Dyskinesia (PCD)
Acronym: LuFu_PCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: Rigshospitalet, Denmark (Other); Hospital Vall d'Hebron (Other); KU Leuven (Other); Amsterdam UMC, location VUmc (Other); University of Valencia (Other); NOVA Medical School (Other); University of Geneva, Switzerland (Other); University of Bern (Other); Ruhr University of Bochum (Other); Charite University, Berlin, Germany (Other); Hannover Medical School (Other); Medical University of Vienna (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University College, London (Other); University of Dundee (Other); University of Southampton (Other); University of Leicester (Other); University of Pisa (Other); Federico II University (Other); Bambino Gesù Hospital and Research Institute (Other); University of Nicosia (Other); Oslo University Hospital (Other); Hospital de Niños R. Gutierrez de Buenos Aires (Other); Hacettepe University (Other); Marmara University (Other); University Hospital, Motol (Other); University Children's Hospital, Zurich (Other); The Leeds Teaching Hospitals NHS Trust (Other); Hadassah Medical Organization (Other); Göteborg University (Other); Schneider Children's Medical Center, Israel (Other); University of Sao Paulo (Other); University Hospital of Cologne (Other); University of Belgrade (Other); University Hospital, Martin (Other); Abderrahmane Mami Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JR_Lufu_PCD_01_2020-1
Record Dates: First submitted 2021-01-12; First posted 2021-01-20 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Ciliary Motility Disorders; Primary Ciliary Dyskinesia
MeSH Terms: conditions — Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genetic diagnosis
  Interventions: Genetic: Genetic diagnosis

INTERVENTIONS:
Genetic: Genetic diagnosis — No Intervention foreseen, but genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD and at least one other method confirming PCD-diagnosis is needed

SUMMARY:
Primary Ciliary Dyskinesia (PCD) is a rare genetic disorder characterized by dysfunction of motile cilia associated with recurrent infections of the airways, laterality defects (Situs inversus totalis in about 50% of cases) and fertility problems. At present, mutations in > 45 genes associated with PCD and mucociliary clearance disorders have been identified, representing most likely two thirds of all human cases.

Aim of this study are:

* Correlation between genotype and lung function of patients with genetically confirmed PCD in an international cohort on a longitudinal basis
* Determination of further parameters, such as body mass index (BMI), possibly associated with lung function in genetically confirmed PCD patients

DETAILED DESCRIPTION:
Background Primary Ciliary Dyskinesia (PCD) is a rare genetic disorder characterized by dysfunction of motile cilia associated with recurrent infections of the airways, laterality defects (Situs inversus totalis in about 50% of cases) and fertility problems. At present, mutations in > 40 genes associated with PCD and mucociliary clearance disorders have been identified, representing most likely two thirds of all human cases. While being involved in the majority of identified PCD genes, our working group has a great expertise in genetic analysis and diagnostic work-up of patients with PCD.

Hallmark symptom of PCD is the chronic purulent lung disease due to the reduced mucociliary clearance. Chronic inflammation and recurrent infections of the airways promote continuous lung damage, bronchiectasis and could finally lead to total lung failure. For other congenital diseases with chronic lung conditions, e.g. cystic fibrosis (CF), an affected lung function with a steady decline is well described and spirometry is widely used to monitor disease progression. For PCD there are only limited data available and studies often comprise small cohorts. In general, available data assume a decline of lung function in PCD patients compared to healthy individuals, but less pronounced than in CF. Altogether, results of the studies remain heterogeneous, in particular concerning the influence of an early diagnosis and a proper treatment on lung function.

Furthermore, despite a significant progression in genetically solved cases there are almost no data on genotype specific lung function in patients with PCD. Recently, there are few studies indicating an association between specific ultrastructural or genetic defects, e.g. patients carrying mutations in the genes MCIDAS (Multicilin), CCNO (Cyclin O), CCDC39 (Coiled-Coil Domain Containing 39) and CCDC40 (Coiled-Coil Domain Containing 40) and a severe clinical course in particular a worse respiratory phenotype. There might be a less severe phenotype in PCD sub-types due to mutations in genes encoding radial spoke components.

Currently a systematic review shows the high variation of spirometric indices in a great PCD cohort. These findings underline the great necessity of detailed characterization of genotype specific phenotypes with focus on important parameters such as lung function to better understand the natural history of distinct PCD-variants with a view to improve individual patient care by tailored treatment activity according to likely disease severity.

Aim of this study are:

* Correlation between genotype and lung function of patients with genetically confirmed PCD in an international cohort on a longitudinal basis
* Determination of further parameters, such as body mass index (BMI), possibly associated with lung function in genetically confirmed PCD patients

Inclusion criteria:

* Patients with a genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD and at least one other method confirming PCD-diagnosis
* Children and adults diagnosed with PCD of all age groups and able to perform spirometry
* Longitudinal datasets with measurements of lung function (FEV1 (forced expiratory volume in 1 second), FVC (forced vital capacity), FEV1/FVC, FEF (forced expiratory flow) 25-75) (with date and height at the performed measurement, respectively)
* at least 3-4 different measurements in at least 2 years of follow up are expected - in cases where this is not possible, sporadic data could also be provided
* Delivery of datasets to the international PCD registry (NCT02419365) with all necessary values within the anticipated time schedules

ELIGIBILITY:
* Patients with a genetically confirmed diagnosis of PCD (bi-allelic mutations in a gene, known to cause PCD) with typical clinical symptoms of PCD and at least one other method confirming PCD-diagnosis
* Children and adults diagnosed with PCD of all age groups and able to perform spirometry
* Longitudinal datasets with measurements of lung function (FEV1, FVC, FEV1/FVC, FEF25-75) (with date and height at the performed measurement, respectively) at least 3-4 different measurements in at least 2 years of follow up are expected - in cases where this is not possible, sporadic data could also be provided
* Delivery of datasets to the international PCD registry (14) with all necessary values within the anticipated time schedules

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PCD patients with proven bi-allelic mutations in a gene known to cause PCD
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Genotype-Lungfunction Correlation | up to 20 years (retrospective)
  Lung function (FEV1, FVC, FEF) in correlation to the genetic make-up

CONTACTS AND LOCATIONS:
Overall Officials: Heymut Omran, Prof., MD, Study Chair — University Hospital Muenster
Locations (1):
- University Hospital Münster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided